CLINICAL TRIAL: NCT00042302
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Phase III Study of Tariquidar + Paclitaxel/Carboplatin as First-Line Therapy in Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: TQD LUNG 001
Record Dates: First submitted 2002-07-26; First posted 2002-08-01 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Stage IIIb Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; tariquidar; Paclitaxel; Carboplatin

INTERVENTIONS:
Procedure: Chemotherapy
Drug: tariquidar + paclitaxel/carboplatin
Drug: placebo + paclitaxel/carboplatin

SUMMARY:
To determine whether tariquidar + combined first-line chemotherapy of paclitaxel/carboplatin in patients with Stage IIIb/IV NSCLC will, with an acceptable safety profile, significantly improve overall survival compared with placebo + paclitaxel/carboplatin. To compare the effects of tariquidar/paclitaxel/carboplatin with placebo/paclitaxel/carboplatin on tumor response, time to disease progression, performance status, symptom progression, and quality of life in patients with Stage IIIb/IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have histologically or cytologically proven NSCLC, stage IIIb or stage IV, requiring first-line chemotherapy.
2. Patients who have a WHO performance status of 1 or 0 and life expectancy of greater than 3 months.
3. Patients who are 18 years of age or older and age of consent.
4. Patients who are women of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test (serum or urine) at screening, and must be practicing an adequate method of birth control.
5. Patients who have neutrophils greater or equal to 1.5 x 103/µL; platelets greater or equal to 100 x 103/µL; bilirubin less or equal to 1.5 times the upper limit of normal or less or equal to 26 µmol/L (1.5 mg/dL); transaminases less or equal to 2.5 times the upper limit of normal or, for patients with known liver metastases, less or equal to 5 times the upper limit of normal; and creatinine less or equal to 141 µmol/L (1.6 mg/dL) or calculated creatinine clearance greater or equal to 60 mL/min prior to study treatment.
6. Patients who are able to give written informed consent and comply with the protocol.

Exclusion Criteria:

1. Patients who are eligible for radiotherapy or surgery for curative intent.
2. Patients who have had previous chemotherapy for NSCLC.
3. Patients who have a WHO performance status greater than 1.
4. Patients with bronchoalveolar carcinoma (an adenocarcinoma in which cylindrical tumor cells grow upon the walls of pre-existing alveoli, from WHO histological typing of lung tumors [1]).
5. Patients who have previous or current primary malignancies at other sites within the last 5 years, with the exception of adequately treated cone-biopsied carcinoma of the cervix and basal or squamous cell skin carcinoma.
6. Patients who are a poor medical risk because of other nonmalignant systemic diseases or active uncontrolled infections.
7. Patients who have symptomatic brain metastases.
8. Patients who have peripheral neuropathy of CTC grade 2, 3, or 4.
9. Patients who have other medical or surgical conditions that would contraindicate chemotherapy.
10. Patients who have received experimental therapies within the last 4 weeks.
11. Patients who have known hypervitaminosis or known sensitivity to ascorbic acid, vitamin A, vitamin D, thiamine, riboflavin, pyridoxine, niacinamide, d-panthenol, or vitamin E.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2002-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)